CLINICAL TRIAL: NCT03081871
Title: Design and Testing of a Mobile Cardiovascular Risk Service With Patient Partners
Brief Title: Mobile Cardiovascular Risk Service Trial
Acronym: mCVRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Elizabeth A Chrischilles, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201603819
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases; Personal Health Records; Pharmaceutical Care; Mobile Apps
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web and mobile app access (Experimental): Subjects will have access to both the mobile and web-app versions of the study Personal Health Record to communicate with the study pharmacist and enter and track their health data.
  Interventions: Other: Pharmacist-led cardiovascular risk service (CVRS); Other: Mobile access to study Personal Health Record; Other: Web access to study Personal Health Record
- Web app only access (Active Comparator): Subjects will have access to the web-app version of the study Personal Health Record (and not the mobile app version) to communicate with the study pharmacist and enter and track their health data.
  Interventions: Other: Pharmacist-led cardiovascular risk service (CVRS); Other: Web access to study Personal Health Record

INTERVENTIONS:
Other: Pharmacist-led cardiovascular risk service (CVRS) — CVRS pharmacists will access the study database including patient baseline information obtained from the medical record and patient entered data to make their assessments and recommendations to onsite physicians and onsite clinical pharmacists and individualize their communication with patients. The intervention will provide patient-centered counseling and education to improve medication adherence, lifestyle modifications and/or smoking cessation. The CVRS pharmacist does not make changes to therapy independently but, rather, provides the physicians and on-site pharmacists with action plans and status updates about adherence to Guideline metrics, which should markedly reduce the gaps in guideline-concordant therapy that place patients at risk for CVD events.
Other: Mobile access to study Personal Health Record — Only subjects assigned to the intervention arm will have access to the mobile app version of the study personal Health Record.
  Arms: Web and mobile app access
Other: Web access to study Personal Health Record — Subjects assigned to both the intervention and control arms will have access to the standard website version of the study personal Health Record.

SUMMARY:
Risk factors for cardiovascular disease are poorly controlled even for patients who frequently visit their physician, leading to large numbers of preventable cardiovascular events such as heart attacks and strokes. Research from integrated healthcare systems suggests that risk factors can be controlled better and treatment strategies for cardiovascular disease can be markedly improved by using a centralized cardiovascular risk service (CVRS) managed by pharmacists. The investigators are confident that a pharmacist-managed mHealth CVRS can become a strategy in un-integrated healthcare settings to markedly reduce cardiovascular events in the United States.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) causes 2,200 deaths in Americans every day with one death every 39 seconds. There is evidence that these deaths can be prevented with better risk factor management, however, many risk factors remain uncontrolled. The Patient-Centered Medical Home (Medical Home) which includes self-management, personalized health records and team-based care, has been proposed as a strategy to reduce these gaps in care delivery. Several Cochrane reviews and meta-analyses have found evidence that adding pharmacists to the primary care team improves risk factor control and physician adherence to guidelines. Managed care organizations have found that a centralized cardiovascular risk service (CVRS) managed by pharmacists can reduce mortality. A gap in the literature is that it is not known whether a comprehensive CVRS model would be implemented in typical office practices in un-integrated settings. Simultaneously, systematic reviews of mobile health (mHealth) trials including disease management apps have found no trial that has incorporated communication with a pharmacist and this lack of evidence is a major gap in the mHealth literature.

The objective of this application is to develop and test a mobile app enabled, pharmacist managed CVRS for disseminating and implementing evidence-based guidelines in practice. In addition to developing the app with patients as design partners, the investigators will conduct a multi-center individually randomized study nested within an ongoing NIH trial in medical offices with large geographic, racial and ethnic diversity. The study team will randomize 100 patients from primary care offices to mHealth CVRS (mobile app + web site + pharmacist) or to CVRS only (web site + pharmacist) of whom 55 will be from racial/ethnic minorities. The central hypothesis is that the mHealth CVRS designed with patients as partners will be implemented and significantly improve patient engagement, leading to improved CVD guideline adherence using the Get with The Guidelines and Guideline Advantage metrics. The rationale for this proposed study is that a novel mHealth model that improves secondary prevention of CVD with pharmacist assistance will lead to broader adoption by health systems throughout the US.

The primary Aim is: to examine the feasibility of mHealth technology to disseminate evidence-based risk reduction guidelines in a prospective randomized controlled trial among diverse primary care offices. The investigators postulate that system engagement (primary hypothesis) and adherence to guidelines for secondary prevention of CVD (secondary hypothesis) will be significantly greater in patients randomized to the mHealth intervention compared to the control group.

This study is expected to produce the following outcomes: unique mobile app features that complement the standard CVRS, increased engagement with a CVRS and increased achievement of guideline-concordant therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients age 55 and older;
2. Owns and uses a smartphone;
3. Any ONE of the following guideline-related needs in the past 18 months:

   1. Most recent encounter LDL >= 100 mg/dl
   2. Most recent encounter BP > 140/90 mmHg (or > 150/90 for persons age 60+)
   3. Most recent encounter not taking recommended post-stroke medications
   4. Most recent encounter not taking recommended post-MI medications
   5. Diabetics with most recent encounter not on ACE inhibitor or ARB blocker
   6. Any patient with most recent A1c > 8.0%
   7. Diabetics with no urine microalbumin screening, past 18 months

EXCLUSION CRITERIA:

1. Non-English speaking (app available only in English for this study)
2. No encounter in the past 18 months (they may be receiving care elsewhere and guideline-related needs may not be reliably assessed) at the clinic itself
3. Most recent systolic BP >200 or diastolic BP > 110 mm Hg
4. Any history of significant hepatic disease, including cirrhosis, Hepatitis B or C infection, or laboratory abnormalities (serum ALT or AST > 3 times normal (either AST above 96 U/L or ALT above 99 U/L or total bilirubin > 2.0 mg/dl))
5. History of hemorrhagic stroke
6. Pulmonary hypertension
7. Stage 4 or metastatic cancer
8. Current nursing home residence or has plans to move to one within the next 12 months
9. Has plans to transfer care from the current clinic within the next 6 months
10. Inability to give informed consent or impaired cognitive function
11. Currently pregnant (females only)
12. Currently a prisoner

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Mean number of days on which a patient interacts with the cardiovascular risk service (using either mobile app or web-site) | 4 months post enrollment
  Mean number of days on which a patient interacts with the cardiovascular risk service (using either mobile app or web-site)
Mean number of contacts with a pharmacist | 4 months post enrollment
  Mean number of contacts with a pharmacist

SECONDARY OUTCOMES:
Guideline Adherence score calculated on the subset of guidelines amenable to intervention during the 4 month intervention | 4 months post enrollment
  Guideline Adherence score calculated on the subset of guidelines amenable to intervention during the 4 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Chrischilles, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Siouxland Community Health Center, Sioux City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Public use data sets will be created and made available to other investigators in a timely manner. Data will only be provided in the form of fully HIPAA-de-identified datasets. Data sets will be carefully reviewed to make sure that information such as age and gender cannot be used to gather additional information that could potentially identify individual subjects. All categorical demographic variables will be collapsed into categories large enough so that combinations of demographic categories for age, gender or area of residence will have 10 or more individuals in each cell. The investigators plan to create SAS datasets in transport format and provide data dictionaries describing the contents of each dataset. Investigators requesting access to the data will be asked to complete a data sharing agreement.